CLINICAL TRIAL: NCT04454879
Title: Different Doses of Roxadustat Treatment on Hemoglobin Target-met in Peritoneal Dialysis Patients
Brief Title: Different Doses of Roxadustat Treatment for Anemia in Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Haidian Hospital (Other); Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Dong Jie, Clinical Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Roxadustat，different dose,
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Renal Anemia
Keywords: Roxadustat; renal anemia; Peritoneal Dialysis
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- standard roxadustat dosage group (Experimental): Peritoneal dialysis patients diagnosed with renal anemia will receive standard dosage of roxadustat according to weight.
  Interventions: Drug: Roxadustat
- lower roxadustat dosage group (Experimental): Peritoneal dialysis patients diagnosed with renal anemia will receive lower dosage of roxadustat according to weight.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Patients in the standard dosage group will receive starting dosage of roxadustat 100 mg, three times per week for weight 45-60kg and 120 mg, three times per week for weight greater than 60kg. Patients in the lower dosage group will receive the starting dosage of roxadustat 50 mg, three times per week for weight lower than 50kg, 70 mg, three times per week for weight 50-70kg, 90 mg, three times per week for weight 70-90kg and 110 mg, three times per week for weight 90-110kg, respectively.

SUMMARY:
A multi-center, randomized, controlled study to evaluate the effect of different doses of roxadustate on hemoglobin target-met in peritoneal dialysis patients

DETAILED DESCRIPTION:
Roxadustat is an orally hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI) to promote erythropoiesis on patients with chronic kidney disease. Two phase 3 clinical trials have verified the efficacy and safety of roxadustate as therapy for anemia in patients with CKD and undergoing dialysis. A high increasing rate of Hb or Hb overshooting triggered by roxadustat need dosing reduction or even drug withdrawal, possibly leading to a large Hb variation and adverse subsequences. Therefore, we were of interest to investigate whether a lower starting dose of roxadustat could achieve comparable Hb target at week 12 while lowering the risk for Hb over 130g/L through a prospective peritoneal dialysis (PD) cohort. Peritoneal dialysis patients diagnosed with renal anemia will be divided into standard roxadustat dosage group and lower roxadustat dosage group. After 12 weeks, we will compare the target-met, overshooting and variation ratio of hemoglobin between these two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients diagnosed with Chronic kidney disease stage 5
2. Maintenance on PD for more than three months.
3. Weight between 45Kg and 110Kg
4. Renal anemia, and hemoglobin between 90g/L and 120g/L
5. Stop taking erythropoietin for enough time （erythropoietin treatment discontinuation for ≥3 days if using erythropoietin of 3000U single strength, or ≥7 days if using erythropoietin of 10000U single strength） or free of erythropoietin use
6. Signed the informed consent.
7. Willing to follow the study procedure

Exclusion Criteria:

1. Hematologic malignancy or aplastic anemia.
2. Blood loss or hemolysis.
3. Taking roxadustat, or Allergy or intolerance to roxadustat
4. Severe liver injury or active hepatitis.
5. Pregnancy or breastfeeding
6. Cancer, receiving radiotherapy and chemotherapy within 6 months.
7. Refractory hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
The ratio of hemoglobin achieving the target (115g/L) | 12 weeks
  The ratio of hemoglobin achieving the target (115g/L) on week 8 and week 12.

SECONDARY OUTCOMES:
The variation ratio of hemoglobin | 12 weeks
  The standard deviation of hemoglobin during the follow-up divide by average of hemoglobin
The ratio of hemoglobin over-shooting | 12 weeks
  Hemoglobin higher than 130g/L during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, MD, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Z, Ma T, Xu X, Fu G, Zhao J, Xu Y, Yang B, Song D, Zhu S, Lv J, Dong J. Randomized Study on the Efficacy of Standard Versus Low Roxadustat Dose for Anemia in Patients on Peritoneal Dialysis. Kidney Int Rep. 2021 Dec 27;7(3):455-464. doi: 10.1016/j.ekir.2021.12.025. eCollection 2022 Mar. PMID 35257058